CLINICAL TRIAL: NCT00510809
Title: Safety and Efficacy of Policosanol Monotherapy and When Added to Chronic Statin Therapy: A Pilot Study
Brief Title: Effect of Policosanol as Monotherapy and Adjunctive to Statin Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James Backes, PharmD (Other)
Collaborators: Marcor Development Corporation (Unknown)
Responsible Party: Sponsor-Investigator, James Backes, PharmD, Clinical Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QB840230; 10494
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Results first posted 2012-07-20 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-09

CONDITIONS: High Cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — policosanol; 1-octacosanol; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Policosanol 20mg daily
  Interventions: Drug: Policosanol
- 2 (Placebo Comparator)
  Interventions: Other: Placebo
- 3 (Active Comparator): Policosanol 20mg daily Plus Statin Therapy Already In Use
  Interventions: Drug: Policosanol Plus Already In Use Statin Therapy

INTERVENTIONS:
Drug: Policosanol — Policosanol 20 mg daily
  Other Names: Octacosanol, 1-Octacosanol, N-Octacosanol, Octacosyl Alcohol
  Arms: 1
Other: Placebo — Placebo daily
  Arms: 2
Drug: Policosanol Plus Already In Use Statin Therapy — Policosanol 20 mg daily Statin Therapy
  Other Names: Octacosanol, 1-Octacosanol, N-Octacosanol, Octacosyl Alcohol; Statin
  Arms: 3

SUMMARY:
To determine the effects of policosanol on the cholesterol profile.

DETAILED DESCRIPTION:
The primary objectives of this study are to determine the changes in the lipid profile [LDL-C, HDL-C, triglycerides, total cholesterol] and the emerging risk factor, Lp(a), when policosanol is added to statin therapy. Additionally, one more primary objective is to evaluate the safety of the combination regimen.

ELIGIBILITY:
Inclusion Criteria:

* LDL > 100
* Male or Non-Pregnant Female. Women must be surgically sterile or postmenopausal and not using hormone replacement therapy (HRT) or using a stable, consistent HRT dose with intentions to continue therapy throughout the course of the study
* Mentally competent to understand study rationale and protocol
* Speak and read English
* Currently receiving low to moderate dose statin therapy with plans to continue to the same dose for at least 8 weeks. Low to moderate dose statins include the following daily doses: atorvastatin ≤20 mg, fluvastatin ≤40 mg, lovastatin ≤40 mg, pravastatin ≤40 mg, rosuvastatin ≤10 mg, simvastatin ≤ 40 mg

Exclusion Criteria:

* LDL < 100
* Sensitivity to policosanol
* Currently taking a high-dose statin or other lipid-lowering agents (i.e. high-dose niacin formulations [>500mg/day], bile-acid sequestrants, ezetimibe, fibrates and high-dose Omega-3 fish oils [>900mg of combined EPA/DHA daily])
* Currently taking medications which have the potential to interact with policosanol (i.e. warfarin, high-dose aspirin)
* Active liver disease or ALT level 2.5 times the upper limit of normal
* Chronic disease involving hepatic, renal or coronary artery disease
* Currently experiencing "flu-like" symptoms
* Currently experiencing any form of acute physical injury
* Acute psychiatric disorders
* Immuno-compromised state
* Currently taking systemic steroidal drugs
* Currently pregnant or lactating
* Females of childbearing potential
* Dependence on alcohol or illicit drugs
* Participation in any other clinical trial within the last 30 days
* Displays s/s of acute systemic infection (oral temperature >100°F, WBC>12x10³/µL)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-07; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M. Backes, PharmD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Statin and Policosanol; Statin and Placebo: 20mg daily, double-blind
- Policosanol: 20 mg daily, open label
Period: Overall Study
Arm/Group | Statin and Policosanol | Statin and Placebo | Policosanol
Started | 18 | 18 | 18
Completed | 18 | 18 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Statin and Policosanol | Statin and Placebo | Policosanol | Total
Number analyzed (Participants) | 18 | 18 | 18 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (12) | 54 (14) | 46 (13) | 51 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 9 | 31
  Male | 6 | 8 | 9 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 1 | 4
  White | 18 | 15 | 16 | 49
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 18 | 54

OUTCOME MEASURES:

1. Primary Outcome: Lipid Profile
Time Frame: Change between Week 8 and Baseline
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Statin and Policosanol | Statin and Placebo | Policosanol
Number analyzed (Participants) | 18 | 18 | 18
mg/dl
  Total Cholesterol | -5 (1.67) | -5 (.92) | 2 (1.96)
  LDL-C | -4 (1.95) | 4 (1.49) | 0 (.34)
  HDL-C | 0 (.17) | -1 (.23) | -1 (.39)
  Triglycerides | 4 (1.52) | -2 (3.91) | 35 (4)
  non-HDL | -4 (1.87) | -4 (1.45) | 3 (.53)
  Lp (a) | 0 (.11) | 0 (4.69) | 1 (.08)
  VLDL | -1 (.13) | 1 (.17) | 3 (.1)

2. Secondary Outcome: Adverse Events Reported
Description: All events reported that were deemed to be related, or unrelated, to the study drug.
Time Frame: Week 8
Measure: Number; unit: number of events reported
Arm/Group | Statin and Policosanol | Statin and Placebo | Policosanol
Number analyzed (Participants) | 18 | 18 | 18
number of events reported | 6 | 10 | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the course of the study using subject reports and questionnaires.
Description: Other events include all reported events, whether or not they were deemed to be related to the study drug.
Arm/Group | Statin and Policosanol | Statin and Placebo | Policosanol
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 6/18 | 10/18 | 5/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Statin and Policosanol (N=18) | Statin and Placebo (N=18) | Policosanol (N=18)
Head cold (General disorders) | 2 | 3 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hip pain (General disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Aftertaste (General disorders) | 0 | 1 | 0
Leg cramps (General disorders) | 0 | 1 | 0
Fever (General disorders) | 0 | 1 | 0
Flank pain (General disorders) | 0 | 1 | 0
Breast cancer (Reproductive system and breast disorders) | 1 | 0 | 0
Pulled hamstring (General disorders) | 1 | 0 | 0
constipation (Gastrointestinal disorders) | 1 | 0 | 0
Headache (General disorders) | 1 | 0 | 1
Transient dizziness (General disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes